CLINICAL TRIAL: NCT04725942
Title: Efficacy, Safety and Serum Concentration of Posaconazole Tablets for Prevention of Pulmonary Fungal Infections in Patients With Hematopoietic Stem Cell Transplantation: An Open, Prospective, Observational, Multicenter Cohort Study
Brief Title: Posaconazole for Pulmonary Fungal Infection Prophylaxis in Hematopoietic Stem Cell Transplantation Patients
Status: Completed | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Shanxi Bethune Hospital (Other); The Second Hospital of Hebei Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NI2020003
Record Dates: First submitted 2021-01-12; First posted 2021-01-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Fungal Infection
MeSH Terms: conditions — Lung Diseases, Fungal | interventions — posaconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Oral Posaconazole tablets — Posaconazole tablets (300 mg Q12h D1) taken orally on the day of transplantation, and followed by 300mg Qd, until 90 days after transplantation.

SUMMARY:
This open, prospective, observational multicenter cohort study aims to evaluate the efficacy, safety as well as the effective serum concentration of Posaconazole for prevention of pulmonary fungal infections in patients with hematopoietic stem cell transplantation. The correlation of UGT1A4*3 genotype and Cmin of Posaconazole, as well as invasive fungal disease (IFD) breakthrough rates will be utilized to evaluate the efficacy while the safety of Posaconazole will be assessed by the overall incidence and severity of adverse events in patients.

DETAILED DESCRIPTION:
This open, prospective, observational multicenter cohort study aims to study the efficacy, safety and effective concentration of Posaconazole tablets for prevention of pulmonary fungal infection in patients with hematopoietic stem cell transplantation. A total of 360 hematopoietic stem cell transplantation patients receiving Posaconazole tablets are expected to be enrolled. Posaconazole tablets will be taken orally from the day of transplantation (300 mg Q12h D1) followed by 300 mg Qd, until 90 days after transplantation. The total duration of the study is estimated to be 24 months, with each patient participating for an estimated 3 months. The relationships between UGT1A4*3 genotype and drug serum concentration, IFD incidence, Aspergillus infection rate, IFD-related mortality rate, IFD-free survival rate, and overall survival rate will be used to evaluate the effectiveness of Posaconazole tablets in preventing invasive pulmonary fungal infection in patients with hematopoietic stem cell transplantation. Safety of Posaconazole tablet will be validated by the overall incidence and severity of adverse events in patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 13 years old
* The primary causes of hematopoietic stem cell transplantation include aplastic anemia, acute myeloid leukemia, acute lymphoblastic leukemia, non-Hodgkin's lymphoma, or other hematologic diseases in patients pretreated for hematopoietic stem cell transplantation. The types of transplantation include autologous transplantation, syngeneic transplantation, matched sibling donor transplantation, unrelated donor transplantation and haploidentical transplantation
* The patients themselves or their authorized clients agree to participate in the clinical study and sign the informed consent

Exclusion Criteria:

* Those with evidence of active fungal infection within 3 weeks prior to enrollment
* Allergic to azole drugs
* Severe abnormal liver function
* Rifampicin, isoniazid, phenytoin, carbamazepine, and long-acting barbiturates were used in combination during the study
* Any predictably increased patient risk or other factors that might interfere with the outcome of a clinical trial

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hematopoietic stem cell transplant patients treated with Posaconazole tablets
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
UGT1A4*3 genotype and plasma concentration of posaconazole | From day 0 to day 22
  Blood samples were drawn at baseline (day 0) for analysis of patients' UGT1A4*3 genotypes and assigned to homozygous, wild-type, and heterozygous genotypes. For posaconazole serum concentrations, blood samples were collected at day 0, 4, 8, 15 and 22.

SECONDARY OUTCOMES:
The incidence of invasive fungal disease (IFD) and the incidence of Aspergillus infection | 90 days posaconazole prophylaxis and 7 days after prophylaxis ending
  Patients who developed invasive fungal infections, aspergillus infections or death related with IFD infections during posaconazole prophylaxis treatment were recorded in accordance with IFD diagnostic guidelines (Revision and Update of the Consensus Definitions of Invasive Fungal Disease From the European Organization for Research and Treatment of Cancer and the Mycoses Study Group Education and Research Consortium. Clin Infect Dis. 2020 Sep 12;71(6):1367-1376).
Plasma concentration of the patients who received different dosages of posaconazole as prophylaxis at different time points | Day 0, 4, 8, 15 and 22
  Blood samples were drawn from patients at day 0, 4, 8, 15, and 22 after receiving posaconazole.
The influence of other combined medications for posaconazole plasma concentrations | Duration of 90-day posaconazole prophylaxis
  Blood samples were drawn at day 0, 4, 8, 15 and 22 after receiving posaconazole, while all combined medications during posaconazole prophylaxis were recorded and IFD cases were monitored during the study period.
Effect of GVHD grading on absorption and utilization of posaconazole tablets (plasma concentration) | Duration of 90-day posaconazole prophylaxis
  Gastrointestinal GVHD grades (I-IV) were recorded according to patient symptoms and posaconazole plasma concentrations were measured using blood samples of each patient after receiving posaconazole tablets at day 0, 4, 8, 15 and 22.
Effect of diarrhea on absorption and utilization of posaconazole tablets (plasma concentration) | Duration of 90-day posaconazole prophylaxis
  Diarrhea (acute watery diarrhea, acute hemorrhagic diarrhea, persistent diarrhea, and diarrhea with severe malnutrition) was recorded according to patient symptoms, and posaconazole plasma concentrations were measured using blood samples of each patient after receiving posaconazole tablets at day 0, 4, 8, 15 and 22.
Number/Proportion of patients with immunosuppressive agent application and adjustments | Duration of 90-day posaconazole prophylaxis
  Recording of the number/proportion of patients who received immunosuppressive agents or adjustments of agents.
Measurement and record of neutrophil counts | Duration of 90-day posaconazole prophylaxis
  Measurement of neutrophils in blood samples of patients.
Measurement and record of duration of neutropenia | Duration of 90-day posaconazole prophylaxis
  Measurement of duration of neutropenia in blood samples of patients.
Adverse events | Duration of 90-day posaconazole prophylaxis
  Record of the number, incidence and frequency of adverse events (AE) during the study period and judge whether the AE is drug related, serious, or special interest AE. AE severity is determined according to MedDRA v23.1.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Second Hospital of Hebei Medical University, Shijia Zhuang
  - Shanxi Bethune Hospital, Taiyuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin